CLINICAL TRIAL: NCT00247793
Title: The Effect of Pre- and Postoperative Supplemental Enteral Nutrition in High-Risk Patients Undergoing Elective Cardiac Surgery. A Prospective Double Blind Study.
Brief Title: Immunonutrition in Cardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 96.17.066; Mec 95/232
Record Dates: First submitted 2005-11-01; First posted 2005-11-02 (Estimated); Last update posted 2005-11-02 (Estimated); Status verified 2005-11

CONDITIONS: Thoracic Surgery; Cardiac Surgery; Cardiopulmonary Bypass
Keywords: immunonutrition; preoperative optimization; preoperative enteral nutritional supplement; high risk; cardiac surgery; arginine; omega-3 polyunsaturated fatty acids; nucleotides; glycine; immune enhancing nutritional supplement; immune enhancing formula

INTERVENTIONS:
Drug: Oral Impact (preoperative enteral nutritional supplement)

SUMMARY:
Effect of two preoperative oral immune-enhancing nutritional supplements in patients at high risk of infection after cardiac surgery: a randomized placebo-controlled study.

Introduction: In our first study we showed that the use of a preoperative oral immune-enhancing nutritional supplement (OIENS) resulted in an improved patients' host-defence with a reduction in postoperative infectious morbidity in 'high-risk' cardiac surgery patients. The use of the OIENS resulted also in less postoperative organ dysfunction. Experimental studies have shown that additional glycine results in less ischemia-reperfusion damage and that glycine has anti-inflammatory properties.

Objective: The use of an OIENS in the preoperative period in patients at high risk of infection after elective cardiac surgery with the use of cardiopulmonary bypass (CPB) results in a reduction in infections as in our first study. The addition of 9.6 gram glycine per sachet OIENS results in a further reduction in postoperative dysfunction.

Design: A prospective randomized placebo controlled study with two oral immune enhancing nutritional formula's and an isocaloric control formula. Patients: Seventy-four consecutive patients undergoing cardiac surgery with the use of an CPB who met one or more of the following inclusion criteria: Age 70 years or older, mitral valve replacement or cardiac ejection fraction less then 40%. Exclusion criteria were age < 18 years, proven malignancy, use of corticosteroids, severe renal and liver failure. Definition of a protocol violation was the intake of less then 5 L or more then 10 L of the nutritional supplement in the preoperative period.

Intervention: Patients were split up in three groups by concealed randomisation. One group received the arginine, omega3-PUFAs and nucleotides enriched formula (OIENS). Another group received the OIENS further enriched with glycine (OIENS+glyc). The control group received an isocaloric nutritional supplement without the enrichments.

DETAILED DESCRIPTION:
Objective To study the effect of two preoperative immune enhancing nutritional supplements compared with a control nutritional supplement in 'high risk' risk cardiac surgery patients

Introduction: Elderly patients and patients with a poor ventricular function undergoing cardiac operations with hypothermic cardiopulmonary bypass (CPB), have an increased postoperative morbidity and mortality. Host defence may be diminished due to nutritional deficiencies, hypoperfusion, anaesthesia and operative trauma. Immune function is additionally depressed by the use of CPB and hypothermia. It has been suggested that L-arginine can improve postoperative outcome in cardiac surgery patients, glycine may have a role in protecting tissues against insults such as ischemia-reperfusion and hypoxia, and omega-3 polyunsaturated fatty acids (omega3-PUFA's) can limit the postoperative generalised inflammatory response.

Experimental studies have shown that the use of nutritional supplements containing L-arginine, omega3-PUFA's or nucleotides, boost immune responsiveness after surgery or trauma. L-arginine is a semi-essential amino acid and precursor of nitrous oxide (NO), the most important endothelial vasodilator. In experimental studies, L-arginine improved wound healing, restored postoperative depressed macrophage function and lymphocyte responsiveness and augmented resistance to infections. Arginine protected against ischemia-reperfusion injury by increasing oxygen delivery upon reflow, thereby improving cardiac function. The intake of additional omega3-PUFA's alters cell membrane phospholipid content and prostaglandin synthesis. This might be an important factor in limiting the generalised inflammatory response and subsequent immunosuppression and capillary leakage following major surgery. Purines and pyrimidines are essential nutrients for rapidly dividing cells. The administration of nucleotides in the form of yeast-RNA has improved the host immune response to an infectious challenge. In experimental studies glycine has been proven cytoprotective in stomach, kidney, liver and cardiovascular system. The metabolic response to oral glycine is that it facilitates the uptake op glucose from the circulation.

The immunonutrients, arginine, omega3-PUFA's and yeast-RNA, have been combined into a single oral immune enhancing nutritional supplement (OIENS). In cancer surgery, trauma and critically ill patients 'post event' nutrition with this immune enhancing formula has improved immunocompetence, reduced infections and shortened length of stay in the hospital (LOSH). The onset of the effect of postoperative immune enhancing nutrition starts after 3 days and seems to be dose dependent. For this reason, it can be hypothesised that it may be beneficial to commence an oral immune enhancing nutritional supplement (OIENS) before surgery. A recent published clinical trail showed that the OIENS with these three immunonutrients in high risk cardiac surgery patients improves preoperative clinical relevant immunological parameters, reduced postoperative infectious morbidity and attenuated postoperative organ dysfunction. Recently, the three immunonutrients have been combined with glycine into a new single OIENS. Aim of the present study in 'high risk' cardiac surgery patients was to determine whether the intake of the new OIENS for minimally five days improves preoperative host defence and subsequently reduces postoperative infections and organ dysfunction.

Study design: A prospective randomized placebo-controlled three armed double blind study

Setting: Departments of cardiopulmonary surgery, anesthesiology and intensive care of the Academic Medical Center, Amsterdam, The Netherlands

Patients: Eligible patients will be included in the study after obtaining written informed consent Inclusion criteria: Patients who met one or more of the inclusion criteria: aged 70 years or more, undergoing cardiac surgery with the use of CPB, or patients with a poor left ventricular function (Ejection fraction < 0.40) or patients undergoing a mitral valve replacement.

Exclusion criteria: Age < 21 years, pregnancy, insulin dependent diabetes mellitus, hepatic cirrhosis, known malignancy, the use of chemotherapy, NSAIDs (excluding acetyl salic acid) or corticosteroids, schizophrenia, severe renal insufficiency (creatinine clearance < 25 mL/h), patients with an organ transplantation in the past

Randomization: 74 patients will be randomized by closed envelop method

Intervention: All patients will receive one of the three enteral nutritional supplements. A formula enriched with arginine, omega-3 PUFA's and nucleotides or the enriched formula further enriched with additional glycine or a control formula. Patients that needs postoperative enteral nutritional support will receive the same formula as preoperative. Patients that need no postoperative enteral nutrition nasogastric tube feeding will not receive the nutritional supplement

Endpoints: Patient compliance, infections, postperfusion phenomena, post-operative organ function (need of postoperative support e.g. inotropic, vasopressor support, fluids, myocardial infarction, ventilation parameters, renal function) time of recovery, mortality

ELIGIBILITY:
Inclusion Criteria:

Patients undergoing cardiac surgery with the use of cardiopulmonary bypass, who met one of the following criteria

* age >= 70 years
* poor left ventricular function (ejection fraction < 0.4)
* mitral valve replacement

Exclusion Criteria:

* Age =< 21 years
* Pregnancy
* Insulin dependent diabetes mellitus
* Hepatic Cirrhosis
* Known malignancy
* Use of chemotherapy, NSAIDs (except ASA), or corticosteroids
* Schizophrenia
* Severe renal failure (creatinine clearance < 25 mL/h) before study entrance
* Patients with an organ transplantation in the past

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1996-07; Study Completion 1998-12

PRIMARY OUTCOMES:
Postoperative infectious morbidity
Mortality

SECONDARY OUTCOMES:
Immunological measurements
Postoperative organ function/support
Recovery (Length of ICU stay, postoperative length of hospital stay)

CONTACTS AND LOCATIONS:
Overall Officials: Leon Eijsman, MD, PhD, Principal Investigator — Director department of cardiopulmonary surgery
Locations (1):
- Cardiopulmonary Surgery, Academic Medical Center, Amsterdam, North Holland, Netherlands

REFERENCES:
- [Background] Tepaske R, Velthuis H, Oudemans-van Straaten HM, Heisterkamp SH, van Deventer SJ, Ince C, Eysman L, Kesecioglu J. Effect of preoperative oral immune-enhancing nutritional supplement on patients at high risk of infection after cardiac surgery: a randomised placebo-controlled trial. Lancet. 2001 Sep 1;358(9283):696-701. doi: 10.1016/s0140-6736(01)05836-6. PMID 11551575
- [Background] Higgins TL, Estafanous FG, Loop FD, Beck GJ, Blum JM, Paranandi L. Stratification of morbidity and mortality outcome by preoperative risk factors in coronary artery bypass patients. A clinical severity score. JAMA. 1992 May 6;267(17):2344-8. PMID 1564774
- [Background] Kress HG, Scheidewig C, Schmidt H, Silber R. Reduced incidence of postoperative infection after intravenous administration of an immunoglobulin A- and immunoglobulin M-enriched preparation in anergic patients undergoing cardiac surgery. Crit Care Med. 1999 Jul;27(7):1281-7. doi: 10.1097/00003246-199907000-00011. PMID 10446821
- [Background] Weimann A, Bastian L, Bischoff WE, Grotz M, Hansel M, Lotz J, Trautwein C, Tusch G, Schlitt HJ, Regel G. Influence of arginine, omega-3 fatty acids and nucleotide-supplemented enteral support on systemic inflammatory response syndrome and multiple organ failure in patients after severe trauma. Nutrition. 1998 Feb;14(2):165-72. doi: 10.1016/s0899-9007(97)00429-2. PMID 9530643
- [Background] O'Leary MJ, Coakley JH. Nutrition and immunonutrition. Br J Anaesth. 1996 Jul;77(1):118-27. doi: 10.1093/bja/77.1.118. No abstract available. PMID 8703621
- [Background] Kirk SJ, Barbul A. Role of arginine in trauma, sepsis, and immunity. JPEN J Parenter Enteral Nutr. 1990 Sep-Oct;14(5 Suppl):226S-229S. doi: 10.1177/014860719001400514. No abstract available. PMID 2232107
- [Background] Engelman DT, Watanabe M, Maulik N, Cordis GA, Engelman RM, Rousou JA, Flack JE 3rd, Deaton DW, Das DK. L-arginine reduces endothelial inflammation and myocardial stunning during ischemia/reperfusion. Ann Thorac Surg. 1995 Nov;60(5):1275-81. doi: 10.1016/0003-4975(95)00614-Q. PMID 8526612
- [Background] Sato H, Zhao ZQ, McGee DS, Williams MW, Hammon JW Jr, Vinten-Johansen J. Supplemental L-arginine during cardioplegic arrest and reperfusion avoids regional postischemic injury. J Thorac Cardiovasc Surg. 1995 Aug;110(2):302-14. doi: 10.1016/S0022-5223(95)70226-1. PMID 7543634
- [Background] Jones SM, Thurman RG. L-arginine minimizes reperfusion injury in a low-flow, reflow model of liver perfusion. Hepatology. 1996 Jul;24(1):163-8. doi: 10.1002/hep.510240127. PMID 8707257
- [Background] Nonami Y. The role of nitric oxide in cardiac surgery. Surg Today. 1997;27(7):583-92. doi: 10.1007/BF02388212. PMID 9306558
- [Background] Daly JM, Weintraub FN, Shou J, Rosato EF, Lucia M. Enteral nutrition during multimodality therapy in upper gastrointestinal cancer patients. Ann Surg. 1995 Apr;221(4):327-38. doi: 10.1097/00000658-199504000-00002. PMID 7726669
- [Background] Zhong Z, Thurman RG. A fish oil diet minimizes hepatic reperfusion injury in the low-flow, reflow liver perfusion model. Hepatology. 1995 Sep;22(3):929-35. PMID 7657301
- [Background] Kulkarni AD, Rudolph FB, Van Buren CT. The role of dietary sources of nucleotides in immune function: a review. J Nutr. 1994 Aug;124(8 Suppl):1442S-1446S. doi: 10.1093/jn/124.suppl_8.1442S. PMID 8064400
- [Background] Heyland DK, Novak F, Drover JW, Jain M, Su X, Suchner U. Should immunonutrition become routine in critically ill patients? A systematic review of the evidence. JAMA. 2001 Aug 22-29;286(8):944-53. doi: 10.1001/jama.286.8.944. PMID 11509059
- [Background] Farreras N, Artigas V, Cardona D, Rius X, Trias M, Gonzalez JA. Effect of early postoperative enteral immunonutrition on wound healing in patients undergoing surgery for gastric cancer. Clin Nutr. 2005 Feb;24(1):55-65. doi: 10.1016/j.clnu.2004.07.002. PMID 15681102
- [Background] Hall JC. Glycine. JPEN J Parenter Enteral Nutr. 1998 Nov-Dec;22(6):393-8. doi: 10.1177/0148607198022006393. PMID 9829614
- [Background] Garner JS. The CDC Hospital Infection Control Practices Advisory Committee. Am J Infect Control. 1993 Jun;21(3):160-2. doi: 10.1016/0196-6553(93)90009-s. No abstract available. PMID 8393635
- [Background] Takala J, Uusaro A, Parviainen I, Ruokonen E. Lactate metabolism and regional lactate exchange after cardiac surgery. New Horiz. 1996 Nov;4(4):483-92. PMID 8968981
- [Background] Kaplan LJ, McPartland K, Santora TA, Trooskin SZ. Start with a subjective assessment of skin temperature to identify hypoperfusion in intensive care unit patients. J Trauma. 2001 Apr;50(4):620-7; discussion 627-8. doi: 10.1097/00005373-200104000-00005. PMID 11303155
- [Background] De Backer D, Creteur J, Vincent JL. Perioperative optimization and right heart catheterization: what technique in which patient? Crit Care. 2003 Jun;7(3):201-2. doi: 10.1186/cc2177. Epub 2003 Mar 14. PMID 12793863
- [Background] Davies SJ, Wilson RJ. Preoperative optimization of the high-risk surgical patient. Br J Anaesth. 2004 Jul;93(1):121-8. doi: 10.1093/bja/aeh164. Epub 2004 Apr 30. No abstract available. PMID 15121729
- [Background] Flancbaum L, Ziegler DW, Choban PS. Preoperative intensive care unit admission and hemodynamic monitoring in patients scheduled for major elective noncardiac surgery: a retrospective review of 95 patients. J Cardiothorac Vasc Anesth. 1998 Feb;12(1):3-9. doi: 10.1016/s1053-0770(98)90047-7. PMID 9509349
- [Background] Zhong Z, Wheeler MD, Li X, Froh M, Schemmer P, Yin M, Bunzendaul H, Bradford B, Lemasters JJ. L-Glycine: a novel antiinflammatory, immunomodulatory, and cytoprotective agent. Curr Opin Clin Nutr Metab Care. 2003 Mar;6(2):229-40. doi: 10.1097/00075197-200303000-00013. PMID 12589194
- [Background] MacFie J, Woodcock NP, Palmer MD, Walker A, Townsend S, Mitchell CJ. Oral dietary supplements in pre- and postoperative surgical patients: a prospective and randomized clinical trial. Nutrition. 2000 Sep;16(9):723-8. doi: 10.1016/s0899-9007(00)00377-4. PMID 10978851
- [Background] Beale RJ, Schneider H, Sorensen f, Smithies MN, Bennet ED, Bihari DJ. A multicentre randomised, controlled trial comparing enteral feeding with IMPACT versus IMPACT with Glycine. Intensive Care Medicine 26(suppl 3):S300,2000
- [Background] Weyandt D. Nutritional supplementation after cardiac surgery. Lancet. 2002 Jan 19;359(9302):256; author reply 257-8. doi: 10.1016/S0140-6736(02)07413-5. No abstract available. PMID 11812582
- [Background] Kollef MH, Sharpless L, Vlasnik J, Pasque C, Murphy D, Fraser VJ. The impact of nosocomial infections on patient outcomes following cardiac surgery. Chest. 1997 Sep;112(3):666-75. doi: 10.1378/chest.112.3.666. PMID 9315799
- [Background] Rebollo MH, Bernal JM, Llorca J, Rabasa JM, Revuelta JM. Nosocomial infections in patients having cardiovascular operations: a multivariate analysis of risk factors. J Thorac Cardiovasc Surg. 1996 Oct;112(4):908-13. doi: 10.1016/S0022-5223(96)70090-9. PMID 8873716
- [Background] Fernandez J, Chen C, Anolik G, Brdlik OB, Laub GW, Anderson WA, McGrath LB. Perioperative risk factors affecting hospital stay and hospital costs in open heart surgery for patients > or = 65 years old. Eur J Cardiothorac Surg. 1997 Jun;11(6):1133-40. doi: 10.1016/s1010-7940(97)01216-5. PMID 9237599
- [Background] Heller AR, Fischer S, Rossel T, Geiger S, Siegert G, Ragaller M, Zimmermann T, Koch T. Impact of n-3 fatty acid supplemented parenteral nutrition on haemostasis patterns after major abdominal surgery. Br J Nutr. 2002 Jan;87 Suppl 1:S95-101. doi: 10.1079/bjn2001462. PMID 11895160
- [Background] Vanschoonbeek K, de Maat MP, Heemskerk JW. Fish oil consumption and reduction of arterial disease. J Nutr. 2003 Mar;133(3):657-60. doi: 10.1093/jn/133.3.657. PMID 12612132
- [Background] Kendall SJ, Weir J, Aspinall R, Henderson D, Rosson J. Erythrocyte transfusion causes immunosuppression after total hip replacement. Clin Orthop Relat Res. 2000 Dec;(381):145-55. doi: 10.1097/00003086-200012000-00018. PMID 11127651
- [Background] Shorr AF, Jackson WL, Kelly KM, Fu M, Kollef MH. Transfusion practice and blood stream infections in critically ill patients. Chest. 2005 May;127(5):1722-8. doi: 10.1378/chest.127.5.1722. PMID 15888852
- [Background] Gessler P, Pfenninger J, Pfammatter JP, Carrel T, Dahinden C. Inflammatory response of neutrophil granulocytes and monocytes after cardiopulmonary bypass in pediatric cardiac surgery. Intensive Care Med. 2002 Dec;28(12):1786-91. doi: 10.1007/s00134-002-1525-x. Epub 2002 Oct 17. PMID 12447524
- [Background] Niessen HW, Lagrand WK, Visser CA, Meijer CJ, Hack CE. Upregulation of ICAM-1 on cardiomyocytes in jeopardized human myocardium during infarction. Cardiovasc Res. 1999 Mar;41(3):603-10. doi: 10.1016/s0008-6363(98)00236-3. PMID 10435032
- [Background] Bozzetti F, Braga M, Gianotti L, Gavazzi C, Mariani L. Postoperative enteral versus parenteral nutrition in malnourished patients with gastrointestinal cancer: a randomised multicentre trial. Lancet. 2001 Nov 3;358(9292):1487-92. doi: 10.1016/S0140-6736(01)06578-3. PMID 11705560
- [Background] Setty S, Tune JD, Downey HF. Nitric oxide contributes to oxygen demand-supply balance in hypoperfused right ventricle. Cardiovasc Res. 2004 Dec 1;64(3):431-6. doi: 10.1016/j.cardiores.2004.07.021. PMID 15537496
- [Background] Kubes P, Granger DN. Nitric oxide modulates microvascular permeability. Am J Physiol. 1992 Feb;262(2 Pt 2):H611-5. doi: 10.1152/ajpheart.1992.262.2.H611. PMID 1539722
- [Background] Braga M, Gianotti L, Cestari A, Vignali A, Pellegatta F, Dolci A, Di Carlo V. Gut function and immune and inflammatory responses in patients perioperatively fed with supplemented enteral formulas. Arch Surg. 1996 Dec;131(12):1257-64; discussion 1264-5. doi: 10.1001/archsurg.1996.01430240011001. PMID 8956766
- [Background] Luiking YC, Poeze M, Dejong CH, Ramsay G, Deutz NE. Sepsis: an arginine deficiency state? Crit Care Med. 2004 Oct;32(10):2135-45. doi: 10.1097/01.ccm.0000142939.81045.a0. PMID 15483426
- [Derived] Tepaske R, te Velthuis H, Oudemans-van Straaten HM, Bossuyt PM, Schultz MJ, Eijsman L, Vroom M. Glycine does not add to the beneficial effects of perioperative oral immune-enhancing nutrition supplements in high-risk cardiac surgery patients. JPEN J Parenter Enteral Nutr. 2007 May-Jun;31(3):173-80. doi: 10.1177/0148607107031003173. PMID 17463141